CLINICAL TRIAL: NCT07347093
Title: Reversal of Roux-en-Y Gastric Bypass: A Swedish National Cohort Study
Status: Active, not recruiting | Type: Observational
Sponsor: Vrinnevi Hospital (Other)
Responsible Party: Principal Investigator, Ellen Andersson, Associate professor, senior consultant, Vrinnevi Hospital
Other Study IDs: Dnr 2022-01827-01
Record Dates: First submitted 2025-12-16; First posted 2026-01-16 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Gastric Bypass Surgery; Revisional Bariatric Surgery; Complications After Bariatric Surgery
Keywords: Roux-en-Y gastric bypass; Anatomical reversal; Indications; Complications; Outcomes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults (≥ 18years) who underwent reversal of RYGB: Included patients were adults (≥ 18years) who underwent reversal of RYGB between 2007 and 2023. Exclusion criteria included emergency reversal due to bowel ischemia, reversal following other bariatric procedures (e.g. gastric banding), or partial/functional reversals (e.g., gastro-gastric fistula or anastomosis between the Roux-limb and gastric remnant, without full reversal of RYGB)

SUMMARY:
Objective:

To investigates incidence, indications, symptom relief, complications, and weight outcomes after Roux-en-Y gastric bypass (RYGB) reversal.

Background:

RYGB is an effective treatment for obesity, but in rare cases may be associated with severe long-term complications requiring RYGB reversal. Evidence on incidence and outcomes is limited.

Methods:

This nationwide, multi-center, retrospective cohort study included all patients undergoing RYGB reversal in Sweden between 2007 and 2023. Data were obtained from the Scandinavian Obesity Surgery Registry (SOReg) and medical records.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18years) who underwent reversal of RYGB between 2007 and 2023.

Exclusion Criteria:

* Emergency reversal due to bowel ischemia
* Reversal following other bariatric procedures (e.g. gastric banding)
* Partial/functional reversals (e.g., gastro-gastric fistula or anastomosis between the Roux-limb and gastric remnant, without full reversal of RYGB)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: National registry-based cohort
Sampling Method: Non-Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Symptom relief | Through study completion, an average of 2 years.
  Symptom relief is classified as no, partial, or complete improvement.
  Complete improvement was defined as full resolution of the index symptom (e.g., cessation of hypoglycemia, pain-free status without analgesics).
  Partial improvement denoted a clinically meaningful reduction in symptom severity or frequency that did not meet criteria for complete resolution.
  No improvement indicated persistent symptoms.

SECONDARY OUTCOMES:
Indications for surgery | Through study completion, an average of 2 years.
  Indications are categorized as abdominal pain, malnutrition, gastrointestinal symptoms, post-bariatric hypoglycemia, and psychological distress, and reported as number (frequencies).
Weight outcome after surgery | Through study completion, an average of 2 years.
  Weigth [in kilograms] will be reported at baseline (before surgery), at one year follow-up, and two-year follow-up.
Complications | At 30-day follow-up and one-year follow-up after surgery.
  Complications after surgery are registered as any complication and major complication (defined as Clavien-Dindo classification >=3b), presented as number (frequencies).
Height | Through study completion, an average of 2 years
  Height (in meters) will be used to report BMI (in kg/m2).
BMI | Through study completion, an average of 2 years.
  Weight (in kilograms) and height (in meters) will be combined to report BMI (in kg/m2) at baseline (before surgery), at one year follow-up, andat two-year follow-up.

OTHER OUTCOMES:
Surgical technique | Perioperative/periprocedural
  * Surgical approach (laparoscopic or open procedure)
  * Handling of the Roux limb (resection or reconnection)
  * Jejuno-jejunostomy technique (stapled/handsewn)
  * Pyloroplasty/pyloromyotomy (yes/no)
  * Gastro-gastrostomy technique (stapled/handsewn)
  * Blood loss during surgery (ml)
  * Operation time (minutes) -all data presented as number (frequencies)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen A Andersson, MD, Principal Investigator — Department of Surgery, Vrinnevi Hospital, Norrköping, and Department of Biomedical and Clinical Sciences, Linköping University, Linköping, Sweden
Locations (1):
- Vrinnevi Hospital, Norrköping, Sweden

IPD SHARING:
Plan to Share IPD: No
Since reversal of RYGB is a rare procedure the risk of identifying individual patients is considerable even if data are pseudonymized.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-11-01): https://cdn.clinicaltrials.gov/large-docs/93/NCT07347093/Prot_SAP_000.pdf